CLINICAL TRIAL: NCT04093700
Title: Clinical Outcomes of Surgical Repair of the Glenoid Labrum Using an All-Suture Anchor
Brief Title: MDR SureLock All-Suture Anchor
Status: Terminated | Type: Observational
Why Stopped: The Sponsor decided that the CE marking would not be renewed, and therefore there was no longer a need to continue the study as the data was no longer necessary.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-90SM
Record Dates: First submitted 2019-08-22; First posted 2019-09-18 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Shoulder Pain; Shoulder Injuries; Shoulder Disease; Shoulder Pain Chronic; Shoulder Syndrome; Labral Tear, Glenoid
MeSH Terms: conditions — Shoulder Pain; Shoulder Injuries; Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- SureLock All-Suture Anchor: Subjects that have been implanted with the SureLock All-Suture Anchor to repair the glenoid labrum
  Interventions: Device: SureLock All-Suture Anchor

INTERVENTIONS:
Device: SureLock All-Suture Anchor — Subjects that have been implanted with the SureLock All-Suture Anchor to repair the glenoid labrum

SUMMARY:
To report the outcomes of a series of patients with recurrent anterior and/or posterior shoulder instability who underwent surgical repair of the affected labrum using the SureLock all-suture anchor.

DETAILED DESCRIPTION:
Patient-reported outcomes data have been collected among patients undergoing shoulder labrum repair with SureLock all-suture anchors from January 2014 to June 30, 2020. These patients have completed clinical and quality-of-life outcome instruments pre-operatively, and have been stored securely in the OBERD database. Pre-op scores will be compared to post-op scores and analyzed using a one-way ANOVA test with a post-hoc Scheffe procedure.

Patient identifying information will be removed and de-identified codes will be used. Any new prospective data gathered prospectively for the purposes of this study will be entered and stored securely as above.

Data collection forms will consist of the following Patient-Reported Outcome Surveys: WOSI Index, ASES Shoulder Score, and the SF-12.

ELIGIBILITY:
Inclusion Criteria:

* 14 to 45 years of age
* Surgery performed between 1/1/14-12/31/2021
* Recurrent shoulder instability resulting from an isolated anterior and/or posterior glenoid labral tear
* Completed pre-operative data (WOSI, ASES, SF-12)

Exclusion Criteria:

* Diagnosis of concomitant SLAP tear
* Diagnosis of concomitant full-thickness rotator cuff tear
* Greater than 10% loss of glenoid bone
* Greater than 25% humeral head defect
* Prior surgical intervention for the treatment of shoulder instability (in either the affected shoulder or the contralateral shoulder)
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects who underwent glenoid labrum repair with the SureLock all-suture anchors between 1/1/2014 and 12/31/2021.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Device Performance and Benefits assessed through improvements in shoulder function | Out to 1 year post-op
  Patients undergoing isolated anterior or posterior glenoid labrum repair using the SureLock All-Suture Anchor will experience statistically significant improvement in shoulder function assessed through the Western Ontario Shoulder Instability Index (WOSI) outcome measure. The WOSI is a 21-item scale used to measure shoulder related quality of life in patients with symptomatic shoulder instability.
Device Performance and Benefits assessed through improvements in shoulder function | Out to 1 year post-op
  Patients undergoing isolated anterior or posterior glenoid labrum repair using the SureLock All-Suture Anchor will experience statistically significant improvement in shoulder function assessed through the American Shoulder and Elbow Surgeon Score(ASES) outcome measure. The ASES is a condition-specific scale that is intended to measure functional limitations and pain of the shoulder.

SECONDARY OUTCOMES:
Device Benefits assessed through improvements of health-related quality of life. | Out to 1 year post-op
  Patients undergoing isolated anterior or posterior glenoid labrum repair using the SureLock All-Suture Anchor will experience statistically significant improvement of health-related quality of life through the SF-12. The SF-12 is a short survey that is weighted and summed to provide easily interpretable scaled for physical and mental health. The range is from 0-100, 0 being the lowest level of health and 100 indicates the highest level of health.
Device Safety and Performance assessed through the frequency and incidence of revisions, complications and Adverse Events. | Out to 1 year post-op
  The assessment of safety and performance will be evaluated by analyzing implant survivorship. This will be established by recording the incidence and frequency of revisions, complications and Adverse Events. Relation of the events to either implant or instrumentation should be specified.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Health Research Institute, Lutherville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No